CLINICAL TRIAL: NCT06654622
Title: An Exosome-Based Liquid Biopsy Assay to Detect Molecular Residual Disease for the Identification of High-Risk Patients With Stage II-III Colorectal Cancer
Brief Title: Exosome-based Detection of Molecular Residual Disease in Stage II-III Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/CRMRD
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Colo-rectal Cancer; Colorectal Cancer Recurrent
Keywords: Colorectal cancer; Molecular residual disease; Adjuvant chemotherapy; Stage II-III CRC; exosomal miRNA
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Postoperative serum samples will be used to isolate exosomal miRNAs for MRD analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Training Cohort (Recurrence Group): Stage II-III CRC patients who experienced postoperative recurrence (evaluated by miRNA panel).
- Training Cohort (Non-Recurrence Group): Stage II-III CRC patients who did not experience postoperative recurrence (evaluated by miRNA panel).
- Testing Cohort (Recurrence Group): Validation of miRNA panel and EMRATI score in independent stage II-III CRC patients who experienced postoperative recurrence.
- Testing Cohort (Non-Recurrence Group): Validation of miRNA panel and EMRATI score in independent stage II-III CRC patients who did not experience postoperative recurrence.

SUMMARY:
This study aims to establish an exosome-based liquid biopsy signature to detect molecular residual disease (MRD) in stage II-III colorectal cancer (CRC) patients. Identifying patients with MRD after surgery is crucial for selecting appropriate candidates for adjuvant chemotherapy (ACT), allowing for more personalized treatment approaches and potentially improving patient outcomes.

DETAILED DESCRIPTION:
The current standard for treating stage II-III colorectal cancer involves surgical resection, often followed by adjuvant chemotherapy (ACT) for high-risk patients. However, identifying patients who would benefit most from ACT remains challenging. Molecular residual disease (MRD) in these patients is a critical factor in determining the likelihood of recurrence. This study aims to develop an exosome-based liquid biopsy assay using circulating exosomal microRNAs (exo-miRNAs) to predict the presence of MRD in postoperative patients. By analyzing exo-miRNAs from blood samples collected after surgery, the goal is to identify high-risk patients who may benefit from ACT while sparing low-risk patients from unnecessary treatment. A risk-stratification model, termed the exosome-based molecular residual disease prediction for adjuvant chemotherapy induction (EMRATI) score, will be developed to improve ACT decision-making and enhance clinical outcomes for stage II-III CRC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed stage II or III colorectal cancer.
2. Patients who have undergone curative-intent surgery.
3. Patients with no evidence of distant metastasis (stage IV).
4. Patients aged 18 years or older.
5. Patients who provided written informed consent.

Exclusion Criteria:

1. Patients with stage IV cancer or those receiving neoadjuvant therapy.
2. Patients with non-curative resection or requiring urgent surgery.
3. Patients with a follow-up period of fewer than 3 years.
4. Patients with severe comorbidities or who are unable to participate in follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients with stage II-III colorectal cancer who have undergone curative surgery and require assessment for molecular residual disease to determine whether adjuvant chemotherapy is necessary.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Tumor Evaluation (Recurrence) | Follow-up at regular intervals during the first 3 years post-surgery.
  Assessment of tumor recurrence through clinical and imaging evaluations.

SECONDARY OUTCOMES:
Overall Survival (OS) | Patients will be monitored for overall survival for up to 5 years post-surgery.
  Evaluation of the overall survival (OS) of patients, defined as the time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou H, Zhu L, Song J, Wang G, Li P, Li W, Luo P, Sun X, Wu J, Liu Y, Zhu S, Zhang Y. Liquid biopsy at the frontier of detection, prognosis and progression monitoring in colorectal cancer. Mol Cancer. 2022 Mar 25;21(1):86. doi: 10.1186/s12943-022-01556-2. PMID 35337361
- [Background] Ruiz-Banobre J, Roy R, Alustiza Fernandez M, Murcia O, Jover R, Pera M, Balaguer F, Lopez-Lopez R, Goel A. Clinical significance of a microRNA signature for the identification and predicting prognosis in colorectal cancers with mucinous differentiation. Carcinogenesis. 2020 Nov 13;41(11):1498-1506. doi: 10.1093/carcin/bgaa097. PMID 32911537
- [Background] Matsuyama T, Toiyama Y, Ishikawa T, Okugawa Y, Yasuno M, Maurel J, Kinugasa Y, Uetake H, Goel A. A metastasis-associated microRNA-based liquid biopsy signature for risk-stratification in colorectal cancer: a multicenter cohort study. Clin Transl Med. 2022 Dec;12(12):e998. doi: 10.1002/ctm2.998. No abstract available. PMID 36513881
- [Background] Miyazaki K, Wada Y, Okuno K, Murano T, Morine Y, Ikemoto T, Saito Y, Ikematsu H, Kinugasa Y, Shimada M, Goel A. An exosome-based liquid biopsy signature for pre-operative identification of lymph node metastasis in patients with pathological high-risk T1 colorectal cancer. Mol Cancer. 2023 Jan 6;22(1):2. doi: 10.1186/s12943-022-01685-8. PMID 36609320
- [Background] Mo S, Ye L, Wang D, Han L, Zhou S, Wang H, Dai W, Wang Y, Luo W, Wang R, Xu Y, Cai S, Liu R, Wang Z, Cai G. Early Detection of Molecular Residual Disease and Risk Stratification for Stage I to III Colorectal Cancer via Circulating Tumor DNA Methylation. JAMA Oncol. 2023 Jun 1;9(6):770-778. doi: 10.1001/jamaoncol.2023.0425. PMID 37079312
- [Background] Yoshino T, Argiles G, Oki E, Martinelli E, Taniguchi H, Arnold D, Mishima S, Li Y, Smruti BK, Ahn JB, Faud I, Chee CE, Yeh KH, Lin PC, Chua C, Hasbullah HH, Lee MA, Sharma A, Sun Y, Curigliano G, Bando H, Lordick F, Yamanaka T, Tabernero J, Baba E, Cervantes A, Ohtsu A, Peters S, Ishioka C, Pentheroudakis G. Pan-Asian adapted ESMO Clinical Practice Guidelines for the diagnosis treatment and follow-up of patients with localised colon cancer. Ann Oncol. 2021 Dec;32(12):1496-1510. doi: 10.1016/j.annonc.2021.08.1752. Epub 2021 Aug 16. PMID 34411693
- [Background] Montcusi B, Madrid-Gambin F, Marin S, Mayol X, Pascual M, Cascante M, Pozo OJ, Pera M. Circulating Metabolic Markers Identify Patients at Risk for Tumor Recurrence: A Prospective Cohort Study in Colorectal Cancer Surgery. Ann Surg. 2024 Nov 1;280(5):842-849. doi: 10.1097/SLA.0000000000006463. Epub 2024 Aug 1. PMID 39087328
- [Background] Kotani D, Oki E, Nakamura Y, Yukami H, Mishima S, Bando H, Shirasu H, Yamazaki K, Watanabe J, Kotaka M, Hirata K, Akazawa N, Kataoka K, Sharma S, Aushev VN, Aleshin A, Misumi T, Taniguchi H, Takemasa I, Kato T, Mori M, Yoshino T. Molecular residual disease and efficacy of adjuvant chemotherapy in patients with colorectal cancer. Nat Med. 2023 Jan;29(1):127-134. doi: 10.1038/s41591-022-02115-4. Epub 2023 Jan 16. PMID 36646802
- [Background] Tie J, Cohen JD, Lahouel K, Lo SN, Wang Y, Kosmider S, Wong R, Shapiro J, Lee M, Harris S, Khattak A, Burge M, Harris M, Lynam J, Nott L, Day F, Hayes T, McLachlan SA, Lee B, Ptak J, Silliman N, Dobbyn L, Popoli M, Hruban R, Lennon AM, Papadopoulos N, Kinzler KW, Vogelstein B, Tomasetti C, Gibbs P; DYNAMIC Investigators. Circulating Tumor DNA Analysis Guiding Adjuvant Therapy in Stage II Colon Cancer. N Engl J Med. 2022 Jun 16;386(24):2261-2272. doi: 10.1056/NEJMoa2200075. Epub 2022 Jun 4. PMID 35657320
- [Background] Kandimalla R, Gao F, Matsuyama T, Ishikawa T, Uetake H, Takahashi N, Yamada Y, Becerra C, Kopetz S, Wang X, Goel A. Genome-wide Discovery and Identification of a Novel miRNA Signature for Recurrence Prediction in Stage II and III Colorectal Cancer. Clin Cancer Res. 2018 Aug 15;24(16):3867-3877. doi: 10.1158/1078-0432.CCR-17-3236. Epub 2018 Mar 7. PMID 29514841